CLINICAL TRIAL: NCT03116347
Title: Post-Authorization Safety, Tolerability and Immunogenicity Evaluation of HyQvia in Pediatric Subjects With Primary Immunodeficiency Diseases
Brief Title: Post-Authorization Safety, Tolerability and Immunogenicity Evaluation of HyQvia in Pediatric PIDD Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161504; 2016-003438-26 (EudraCT Number)
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-04

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPOCH 1 (Experimental): Ramp up period for participants who were not treated with HyQvia prior to this study
  Interventions: Biological: HYQVIA
- EPOCH 2 (Experimental): Participants who were treated with HyQvia prior to this study, and those who completed the ramp up period (Epoch 1). After one year in Epoch 2, participants with anti-rHuPH20 antibody titer <160 at all time-points during the study will complete the study termination/completion visit at the next possible occasion. Participants with anti-rHuPH20 antibody titer >=160 during the study and/or at the last measurement will continue for an additional two years of HyQvia treatment and observation.
  Interventions: Biological: HYQVIA
- Epoch 3 (Experimental): Safety follow-up for participants whose anti-rHuPH20 antibody titer was >= 160 during Epoch 1 or Epoch 2 and who experience either a related serious adverse event (SAE) or a related severe adverse event (AE)
  Interventions: Biological: KIOVIG; Biological: Cuvitru

INTERVENTIONS:
Biological: HYQVIA — Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase (IGI, 10% with rHuPH20)
  Other Names: IGI 10% with rHuPH20
  Arms: EPOCH 1; EPOCH 2
Biological: KIOVIG — 100 mg/ml solution for Immune Globulin Intravenous Infusion
  Other Names: IGIV 10%; IGI 10%
  Arms: Epoch 3
Biological: Cuvitru — 200 mg/ml solution for Immune Globulin Subcutaneous Injection
  Other Names: IGSC 20%; IGI 20%
  Arms: Epoch 3

SUMMARY:
The purpose of the study is to acquire additional data on safety, tolerability and immunogenicity of HyQvia in pediatric (age two to <18 years) patients with Primary Immunodeficiency Diseases (PIDD)

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a documented diagnosis of a form of primary humoral immunodeficiency involving a defect in antibody formation and requiring gammaglobulin replacement, as defined according to the International Union of Immunological Societies (IUIS) Scientific Committee 2015 prior to enrollment. The diagnosis must be confirmed by the sponsor´s Medical Director prior to first treatment with investigational product (IP) in the study.
2. Participant is at least two and below 18 years of age at the time of screening.
3. Participant has been receiving a consistent dose of Immunoglobulin G (IgG), administered in compliance with the respective product information for a period of at least three months prior to screening. The average minimum pre-study dose over that interval was equivalent to 300 mg/kg body weight (BW)/four weeks and a maximum dose equivalent to 1000 mg/kg BW/4 weeks.
4. Participant has a serum trough level of IgG > 5 g/L at screening.
5. If female of childbearing potential, participant presents with a negative pregnancy test and agrees to employ adequate birth control measures for the duration of the study.
6. Participant /legally authorized representative is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Participant has a known history of or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1/2.
2. Abnormal laboratory values at screening meeting any one of the following criteria (abnormal tests may be repeated once to determine if they are persistent):

   1. Persistent alanine aminotransferase (ALT) and aspartate amino transferase (AST) >2.5 times the upper limit of normal (ULN) for the testing laboratory
   2. Persistent severe neutropenia (defined as an absolute neutrophil count [ANC] ≤ 500/mm^3)
3. Participant has anemia that would preclude phlebotomy for laboratory studies, according to standard practice at the site.
4. Participant has an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following intravenous (IV) immunoglobulin, subcutaneous (SC) immunoglobulin, and/or Immune Serum Globulin (ISG) infusions.
5. Participant has severe immunoglobulin A (IgA) deficiency (< 7.0 mg/dL) with known anti-IgA antibodies and a history of hypersensitivity. .
6. Participant has a known allergy to hyaluronidase.
7. Participant has active infection and is receiving antibiotic therapy for the treatment of infection at the time of screening.
8. Participant has a bleeding disorder or a platelet count < 20,000/μL, or who, in the opinion of the investigator, would be at significant risk of increased bleeding or bruising as a result of SC therapy.
9. Participant has severe dermatitis that would preclude adequate sites for safe product administration in the opinion of the investigator.
10. Participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
11. Participant is a family member or employee of the investigator.
12. If female, participant is pregnant or lactating at the time of enrollment.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (20):
- Czechia (3):
  - Fakultni nemocnice Brno Odd. Detska klinika, Brno
  - Fakultní nemocnice Hradec Králové, Nový Hradec Králové
  - FN v Motole Interni klinika, Prague
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Groupe Hospitalier Pellegrin - Hôpital des Enfants, Bordeaux, Gironde
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - Hospices Civils de Lyon - Hôpitaux Est - IHOP, Lyon
- Greece (3):
  - Agia Sophia Children's Hospital, Athens
  - General Hospital of Thessaloniki Ippokrateio, Thessaloniki
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki
- United St. Istvan and St. Laszlo Hospital, Budapest, Hungary
- Slovakia (2):
  - 1.Detská klinika, Bratislava
  - Univerzitna Nemocnica Klinika detí a dorastu, Martin
- Sweden (2):
  - Queen Silvia Children's Hospital, Gothenburg
  - Dept. of Pediatric Oncology/Hematology/Immunology-Skånes Universitetssjukhus, Lund
- United Kingdom (5):
  - Bristol Royal Hospital for Children, Bristol, Avon
  - Leeds Children's Hospital, Leeds, West Yorkshire
  - Royal Victoria Hospital, Belfast
  - University Hospital of Wales Heath Park Clinical Research Facility, Cardiff
  - The Great North Children's Hospital Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ciznar P, Roderick M, Schneiderova H, Jesenak M, Krivan G, Brodszki N, Jolles S, Atisso C, Fielhauer K, Saeed-Khawaja S, McCoy B, Yel L. fSCIG 10% in pediatric primary immunodeficiency diseases: a European post-authorization safety study. Allergy Asthma Clin Immunol. 2024 Sep 17;20(1):47. doi: 10.1186/s13223-024-00904-9. PMID 39289739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 sites from 30 May 2017 to 15 January 2021. A total of 42 participants were enrolled and treated in this study. This study consisted of 3 treatment periods: Epoch 1, Epoch 2 and Epoch 3. Participant with anti-rHuPH20 antibody titer greater than or equal to (>=) 160 during Epoch 1 or Epoch 2 and who experienced either a related serious adverse event or related severe adverse event were followed to Epoch 3.
Pre-assignment Details: Participants who were treated with HyQvia in Epoch 1 followed by Epoch 2 were referred to as "HyQvia new starters" and participants who started directly in Epoch 2 were referred to as "HyQvia pre-treated". 1 participant from "HyQvia new starters" group discontinued Epoch 2 and entered Epoch 3 due to a severe related adverse event. Participant did not receive HyQvia treatment in Epoch 3. Therefore, no further safety and efficacy data were collected in Epoch 3.
Groups:
- HyQvia New Starters: Participants who were treated with non-HyQvia treatment by time of enrollment were enrolled in Epoch 1 (ramp-up) and treated with HyQvia subcutaneously (SC) with a dose or interval ramp-up period of up to 6 weeks. HyQvia dose was planned to be equivalent to 100% (±5%) of pre-study treatment. Dosage Frequency was one treatment interval of one week, then one treatment interval of two weeks, then one treatment interval of three weeks (for participants in whom treatment was expected to be every four weeks). The ramp-up period was followed by Epoch 2 (no ramp-up) with HyQvia SC treatment at every 3 or 4 weeks, depending on the participant's previous dosing schedule and the discretion of the investigator and participant, for up to 20 months.
- HyQvia Pre-treated: Participants already treated with HYQVIA by the time of enrollment were directly enrolled in Epoch 2 and treated with HyQvia SC at every 3 or 4 weeks for up to 20 months. HyQvia dose was planned to be equivalent to 100% (±5%) of pre-study treatment with a dosage frequency of once every three or four weeks, based on the participants previous dosing schedule and the discretion of the investigator and participant.
Period: Overall Study
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Started | 23 | 19
Started Epoch 1 | 23 | 0
Completed Epoch 1 | 22 | 0
Started Epoch 2 | 22 | 19
Completed Epoch 2 | 22 | 17
Moved From Epoch 2 to Epoch 3 | 1 | 0
Completed Epoch 3 | 1 | 0
Completed | 22 | 17
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants in the full analysis set (enrolled set) who received at least one dose of HyQvia.
Groups:
- HyQvia New Starters: Participants who were treated with non-HyQvia treatment by time of enrollment were enrolled in Epoch 1 (ramp-up) and treated with HyQvia SC with a dose or interval ramp-up period of up to 6 weeks. HyQvia dose was planned to be equivalent to 100% (±5%) of pre-study treatment. Dosage Frequency was one treatment interval of one week, then one treatment interval of two weeks, then one treatment interval of three weeks (for participants in whom treatment was expected to be every four weeks). The ramp-up period was followed by Epoch 2 (no ramp-up) with HyQvia SC treatment at every 3 or 4 weeks, depending on the participant's previous dosing schedule and the discretion of the investigator and participant, for up to 20 months.
- Total: Total of all reporting groups
Arm/Group | HyQvia New Starters | HyQvia Pre-treated | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.3 (3.82) | 11.7 (4.33) | 11 (4.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 19 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 19 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Any Severe Related Treatment-emergent Adverse Events (TEAEs) Per Infusion (Excluding Infections)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant administered an investigational product (IP) that does not necessarily have a causal relationship with the treatment. TEAEs were the AEs with onset after date-time of first dose of IP, or any medical condition present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. TEAEs that were recorded as "possibly related" or "probably related" to HYQVIA were considered HYQVIA-related adverse events. Number of participants with any severe related TEAEs (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 1 | 0

2. Primary Outcome: Safety: Rate of Any Severe Related TEAEs Per Infusion (Excluding Infections)
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. TEAEs were the AEs with onset after date-time of first dose of IP, or any medical condition present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. TEAEs that were recorded as "possibly related" or "probably related" to HYQVIA were considered HYQVIA-related adverse events. Severe related TEAEs rate per infusion was calculated as number of severe related TEAEs/total number of infusions administered to participants in the analysis set. Rate of any severe related TEAEs per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of Severe Related TEAEs/Infusion
Units Other Than Participants: Infusions
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusions) | 464 | 331
Number of Severe Related TEAEs/Infusion | 0.004 | 0

3. Primary Outcome: Safety: Number of Participants With Any Related Serious TEAEs Per Infusion (Excluding Infections)
Description: TEAEs were the AEs with onset after date-time of first dose of IP, or any medical condition present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs that were recorded as "possibly related" or "probably related" to HYQVIA were considered HYQVIA-related adverse events. Number of participants with any related serious TEAEs per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 0 | 0

4. Primary Outcome: Safety: Rate of Any Related Serious TEAEs Per Infusion (Excluding Infections)
Description: TEAEs were the AEs with onset after date-time of first dose of IP, or any medical condition present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in-patient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs that were recorded as "possibly related" or "probably related" to HYQVIA were considered HYQVIA-related adverse events. Rate of related serious TEAEs per infusion was calculated as number of related serious TEAEs/total number of infusions administered to participants in the analysis set. Rate of any related serious TEAEs per Infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of Related Serious TEAEs/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Number of Related Serious TEAEs/Infusion | 0 | 0

5. Secondary Outcome: Efficacy: Change From Baseline in Total Serum Trough Levels of Immunoglobulin G (IgG) at Month 12
Description: Change from baseline in total serum trough levels of IgG in Epoch 1 and 2 was reported. Baseline was defined as the last non-missing value before the initial dose of HYQVIA.
Time Frame: Baseline, Month 12
Population: Full analysis set included all participants who provide informed consent and meet enrollment eligibility. Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 20 | 17
Gram per liter (g/L) | 0.035 (1.6983) | -0.709 (2.6576)

6. Secondary Outcome: Efficacy: Change From Baseline in Serum Trough Levels of IgG Subclasses at Month 12
Description: Change from baseline in Serum trough levels of IgG subclasses 1, 2, 3, and 4 in Epoch 1 and 2 was reported. Baseline was defined as the last non-missing value before the initial dose of HYQVIA.
Time Frame: Baseline, Month 12
Population: All participants in the full analysis set (enrolled set) who received at least one dose of HyQvia. Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 16 | 15
g/L
  IgG Subclass 1 : Changed at Month 12 | -0.813 (1.1087) | -0.467 (1.5976)
  IgG Subclass 2 : Changed at Month 12 | 0.000 (0.8944) | -0.667 (1.3452)
  IgG Subclass 3 : Changed at Month 12 | 0.000 (0.3651) | 0.133 (0.3519)
  IgG Subclass 4 : Changed at Month 12 | 0.094 (0.0854) | -0.027 (0.0799)

7. Secondary Outcome: Efficacy: Change From Baseline in Trough Levels of Specific Antibodies to Clostridium Tetani Toxoid IgG at Month 12
Description: Change from baseline in trough levels of specific antibodies in clostridium tetani toxoid IgG at Month 12 was reported. Baseline was defined as the last non-missing value before the initial dose of HYQVIA. Here, IU/ml was defined as "International units per milliliter".
Time Frame: Baseline, Month 12
Population: All participants in the full analysis set (enrolled set) who received at least one dose of HyQvia. Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure. Specific antibody data were not scheduled to be collected at Epoch 2 Month 0, so for most participants baseline could not be defined and change from baseline was not reported in HYQVIA Pre-treated arm.
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 21 | 0
IU/ml | -0.218 (0.9345) |

8. Secondary Outcome: Efficacy: Change From Baseline in Trough Levels of Specific Antibodies to Hepatitis B Virus (HBV) at Month 12
Description: Change from baseline in trough levels of specific antibodies in HBV at Month 12 was reported. Baseline was defined as the last non-missing value before the initial dose of HYQVIA.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 16 | 0
International units per liter (IU/L) | 167.875 (147.4887) |

9. Secondary Outcome: Efficacy: Change From Baseline in Trough Levels of Specific Antibodies to Haemophilus Influenzae B IgG at Month 12
Description: Change from baseline in trough levels of specific antibodies in Haemophilus influenzae B IgG at Month 12 was reported. Baseline was defined as the last non-missing value before the initial dose of HYQVIA.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Milligram per liter (mg/L)
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 20 | 0
Milligram per liter (mg/L) | -0.017 (0.9503) |

10. Secondary Outcome: Safety: Percentage of Participants Who Achieved a Treatment Interval of Three or Four Weeks in Epoch 2
Description: Percentage of participants who achieved a treatment interval of three or four weeks in Epoch 2 was reported.
Time Frame: Up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Percentage of participants
  Every 3 weeks treatment interval | 39.1 | 15.8
  Every 4 weeks treatment interval | 60.9 | 84.2

11. Secondary Outcome: Safety: Percentage of Participants Who Maintained a Treatment Interval of Three or Four Weeks in Epoch 2 up to 12 Months
Description: Percentage of participants who maintained a treatment interval of three or four weeks in Epoch 2 up to 12 months was reported.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Percentage of participants | 87.0 | 78.9

12. Secondary Outcome: Safety: Number of Participants With Local TEAEs (Excluding Infections)
Description: TEAEs were the AEs with onset after date-time of first dose of IP, or any medical condition present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. Number of Participants with local TEAEs (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 11 | 3

13. Secondary Outcome: Safety: Rate of Local TEAEs Per Infusion (Excluding Infections)
Description: Rate of local TEAEs per infusion was calculated as number of local adverse events/total number of infusions administered to participants in the analysis set. Only events are included which start prior to participants start date of non-response. Rate of local TEAEs per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of local TEAEs/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Number of local TEAEs/Infusion | 0.082 | 0.009

14. Secondary Outcome: Safety: Number of Participants With Local Adverse Reaction (Excluding Infections)
Description: Adverse reaction was defined as any TEAE that meets any of the following criteria: 1) A TEAE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or; 2) A TEAE that begins during infusion of IP or within 72 hours following the end of IP infusion, or; 3) A TEAE for which causality assessment is missing or indeterminate. Number of participants with local adverse reactions (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 11 | 3

15. Secondary Outcome: Safety: Rate of Local Adverse Reaction Per Infusion (Excluding Infections)
Description: Rate of local adverse reaction per infusion was calculated as number of local adverse reaction events/total number of infusions administered to participants in the analysis set. Rate of local adverse reactions per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of Local AR events/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Number of Local AR events/Infusion | 0.080 | 0.009

16. Secondary Outcome: Safety: Number of Participants With Systemic TEAEs (Excluding Infections)
Description: TEAEs were the AEs with onset after date-time of first dose of IP, or any medical condition present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. Number of participants with systemic TEAEs (excluding infections) was reported..
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 15 | 10

17. Secondary Outcome: Safety: Rate of Systemic TEAEs Per Infusion (Excluding Infections)
Description: Rate of systemic TEAEs per infusion was calculated as number of systemic adverse events/total number of infusions administered to participants in the analysis set. Rate of systemic TEAEs per infusion was assessed based on events per infusion.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of systemic TEAEs/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Number of systemic TEAEs/Infusion | 0.138 | 0.142

18. Secondary Outcome: Safety: Number of Participants With Systemic Adverse Reaction (Excluding Infections)
Description: Adverse reaction was defined as any TEAE that meets any of the following criteria: 1) A TEAE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or; 2) A TEAE that begins during infusion of IP or within 72 hours following the end of IP infusion, or; 3) A TEAE for which causality assessment is missing or indeterminate. Number of participants with systemic adverse reaction (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 3 | 1

19. Secondary Outcome: Safety: Rate of Systemic Adverse Reaction Per Infusion (Excluding Infections)
Description: Rate of Systemic adverse reactions per infusion was calculated as number of systemic adverse reaction events/total number of infusions administered to participants in the analysis set. Rate of systemic adverse reactions per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of systemic AR events/Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number of systemic AR events/Infusion | 0.011 | 0.012

20. Secondary Outcome: Safety: Number of Participants With Any TEAEs (Excluding Infections)
Description: TEAEs were the AEs with onset after date-time of first dose of IP, or any medical condition present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. Number of participants with any TEAEs (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 18 | 11

21. Secondary Outcome: Safety: Rate of TEAEs Per Infusion (Excluding Infections)
Description: Rate of TEAEs per infusion was calculated as number of adverse events/total number of infusions administered to participants in the analysis set. Rate of TEAEs per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of TEAEs/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Number of TEAEs/Infusion | 0.220 | 0.151

22. Secondary Outcome: Safety: Number of Participants With Any Adverse Reactions (Excluding Infections)
Description: Adverse reaction was defined as any TEAE that meets any of the following criteria: 1) A TEAE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or; 2) A TEAE that begins during infusion of IP or within 72 hours following the end of IP infusion, or; 3) A TEAE for which causality assessment is missing or indeterminate. Number of participants with any adverse reactions (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 12 | 3

23. Secondary Outcome: Safety: Rate of Any Adverse Reaction Per Infusion (Excluding Infections)
Description: Rate of all adverse reactions per infusion was calculated as number of adverse reaction events/total number of infusions administered to participants in the analysis set. Rate of any adverse reactions per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Adverse reaction event/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Adverse reaction event/Infusion | 0.091 | 0.021

24. Secondary Outcome: Safety: Number of Participants With Any Temporally Associated TEAEs (Excluding Infections)
Description: Temporally-associated TEAEs were defined as TEAEs which begin during infusion of IP or within 72 hours following the end of IP infusion. Number of participants with any temporally associated TEAEs (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 13 | 6

25. Secondary Outcome: Safety: Rate of Any Temporally Associated TEAEs Per Infusion (Excluding Infections)
Description: Rate of any temporally associated TEAEs per infusion was calculated as number of temporally associated adverse events/total number of infusions administered to participants in the analysis set. Temporally-associated TEAEs were defined as TEAEs which begin during infusion of IP or within 72 hours following the end of IP infusion. Rate of any temporally associated TEAEs per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Temporally associated TEAEs/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Temporally associated TEAEs/Infusion | 0.106 | 0.027

26. Secondary Outcome: Safety: Number of Participants With Any Related (Causally) and/or Temporally Associated TEAEs (Excluding Infections)
Description: Number of participants with any related (causally) and/or temporally associated TEAEs (excluding infections) was reported. Temporally-associated TEAEs were defined as TEAEs which begin during infusion of IP or within 72 hours following the end of IP infusion.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 13 | 6

27. Secondary Outcome: Safety: Rate of Any Related (Causally) and/or Temporally Associated TEAEs Per Infusion (Excluding Infections)
Description: Rate of any related (causally) and/or temporally associated TEAEs per infusion was calculated as number of related and/or temporally associated adverse events/ total number of infusions administered to participants in the analysis set. TEAEs recorded in the study database as "possibly related" or "probably related" to HYQVIA are considered HYQVIA-related adverse events. Temporally-associated TEAEs were defined as TEAEs which begin during infusion of IP or within 72 hours following the end of IP infusion. Rate of any related (causally) and/or temporally associated TEAEs per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Related Temporally TEAEs/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Related Temporally TEAEs/Infusion | 0.112 | 0.033

28. Secondary Outcome: Safety: Number of Participants With Any Serious TEAEs (Excluding Infections)
Description: Serious TEAE were the AEs that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in-patient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Number of participants with any serious TEAEs (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants | 0 | 3

29. Secondary Outcome: Safety: Rate of Serious TEAEs Per Infusion (Excluding Infections)
Description: Rate of serious TEAEs per infusion was calculated as number of serious adverse events/total number of infusions administered to participants in the analysis set. Rate of serious TEAEs per infusion (excluding infections) was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Number of serious TEAEs/Infusion
Units Other Than Participants: Infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusion) | 464 | 331
Number of serious TEAEs/Infusion | 0 | 0.012

30. Secondary Outcome: Safety: Number of Participants Who Developed Positive Titer (>=160) of Binding or Neutralizing Antibodies to rHuPH20
Description: Number of participants who developed positive titer (>=160) of binding or neutralizing antibodies to rHuPH20 was reported.
Time Frame: From start of study drug administration up to 20 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Participants
  Participants with positive titer (>=160) of binding antibodies | 0 | 0
  Participants with neutralizing antibodies | 0 | 0

31. Secondary Outcome: Other Analysis: Number of Infusions Per Month
Description: Number of infusions per month was calculated as total number of infusions per duration of treatment (days) * 30.4 days per month.
Time Frame: Up to 20 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Infusion/Month
Units Other Than Participants: Infusions
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusions) | 464 | 331
Infusion/Month | 1.30 [1.1 to 1.7] | 1.20 [1.0 to 1.6]

32. Secondary Outcome: Other Analysis: Number of Infusion Sites (Needle-Sticks) Per Infusion
Description: Number of infusion sites (needle-sticks) per infusion was calculated as total number of infusion sites / total number of infusions. Only infusions with complete data available were included.
Time Frame: Up to 20 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Infusion sites (needle sticks)/Infusion
Units Other Than Participants: infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (infusion) | 464 | 331
Infusion sites (needle sticks)/Infusion | 1.65 (0.442) | 1.25 (0.403)

33. Secondary Outcome: Other Analysis: Number of Infusion Sites (Needle-Sticks) Per Month
Description: Number of infusion sites per month was calculated as total number of infusion sites / duration of treatment (days) * 30.4 days. Only infusions with complete data available were included.
Time Frame: Up to 20 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Infusion sites (needle sticks)/Month
Units Other Than Participants: infusion
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (infusion) | 464 | 331
Infusion sites (needle sticks)/Month | 1.96 (0.780) | 1.33 (0.634)

34. Secondary Outcome: Other Analysis: Duration of Infusion
Description: The duration of infusion was defined as the difference between the end time and the start time of the HyQvia infusion.
Time Frame: From start of study drug administration up to 20 months.
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Minutes
Units Other Than Participants: Infusions
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusions) | 395 | 247
Minutes | 75.0 [10 to 215] | 101.0 [15 to 257]

35. Secondary Outcome: Other Analysis: Maximum Infusion Rate Per Site
Description: Maximum infusion rate per site was reported.
Time Frame: Up to 20 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milliliter per hour per site (mL/h/site)
Units Other Than Participants: Infusions
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusions) | 402 | 265
Milliliter per hour per site (mL/h/site) | 181.54 (77.772) | 171.73 (90.203)

36. Secondary Outcome: Other Analysis: Infusion Volume Per Site
Description: Infusion volume per site was calculated as actual IgG volume (milliliter [mL]) / total number of infusion sites (hour) used.
Time Frame: Up to 20 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milliliter per hour
Units Other Than Participants: Infusions
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusions) | 403 | 286
Milliliter per hour | 112.39 (71.427) | 178.23 (98.523)

37. Secondary Outcome: Other Analysis: Number of Infusions That Were Interrupted or Stopped Due to an AE
Description: Number of infusions that were interrupted or Stopped due to an AE was reported.
Time Frame: Up to 20 months
Population: as for baseline characteristics
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 23 | 19
Number analyzed (Infusions) | 464 | 331
Infusions
  Number of infusions interrupted | 4 | 0
  Number of infusions Stopped | 1 | 0

38. Secondary Outcome: Other Analysis: Number of Weeks to Reach Final 3 or 4-week Dose Interval in Epoch 1
Description: Final dose interval, defined as three or four weeks infusion interval in Epoch 1 of treatment period, was reported.
Time Frame: Up to 20 months
Population: Safety analysis set included all participants in the full analysis set (enrolled set) who received at least one dose of HyQvia. Here, "Overall number of Participants Analyzed" signifies participants who are evaluable for this outcome measure. Data collection and analysis was not planned for HyQvia pre-treated group.
Measure: Median (Full Range); unit: Weeks
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 22 | 0
Weeks | 6.10 [3.0 to 7.0] |

39. Secondary Outcome: Health Related Quality of Life (HR QoL): Change From Baseline in Pediatric Quality of Life Questionnaire (PedsQL)
Description: PedsQL Generic Core Scale (GCS) was used for QOL assessment. It encompasses 4 dimensions (physical functioning [PF], emotional functioning [EF], social functioning [SF], school functioning [ScF]). Age groups are: Toddler (2-4 years), Young child (5-7 years), Child (8-12 years), and Teens (13-<18 years). Depending on the participants age, the questionnaire may be completed by either the participant or the parent/caregiver as appropriate. For the Toddler group, the PedsQL GCS consisted of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL consisted of 23 items, with a 3-point Likert scale (0, 2, 4) for the young child, and a 5-point Likert scale for the child and teens groups. All Scores were transformed on a scale from 0 to 100 where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate better quality of life. A negative change from baseline indicates worse quality of life. Baseline: last non-missing value before the initial dose of HYQVIA.
Time Frame: Baseline up to 20 months
Population: Safety analysis set included all participants in the full analysis set (enrolled set) who received at least one dose of HyQvia. Here, "Overall number of Participants Analyzed" signifies participants who are evaluable for this outcome measure and "Number analyzed" signifies participants who are evaluable for this outcome at specific time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 5 | 8
Score on a scale
  PF in Toddler: Change up to 20 months: number analyzed (Participants) | 0 | 1
  PF in Toddler: Change up to 20 months |  | -3.12 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  PF in Young child: Change up to 20 months: number analyzed (Participants) | 0 | 1
  PF in Young child: Change up to 20 months |  | -31.25 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  PF in Child: Change up to 20 months: number analyzed (Participants) | 2 | 1
  PF in Child: Change up to 20 months | 7.81 (6.626) | -71.88 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  PF in Teens: Change up to 20 months: number analyzed (Participants) | 3 | 5
  PF in Teens: Change up to 20 months | -12.65 (12.726) | 13.75 (24.664)
  EF in Toddler: Change up to 20 months: number analyzed (Participants) | 0 | 1
  EF in Toddler: Change up to 20 months |  | 0.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  EF in Young child: Change up to 20 months: number analyzed (Participants) | 0 | 1
  EF in Young child: Change up to 20 months |  | -25.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  EF in Child: Change up to 20 months: number analyzed (Participants) | 2 | 1
  EF in Child: Change up to 20 months | 5.00 (14.142) | -20.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  EF in Teens: Change up to 20 months: number analyzed (Participants) | 3 | 5
  EF in Teens: Change up to 20 months | -13.33 (7.638) | 1.25 (14.307)
  SF in Toddler: Change up to 20 months: number analyzed (Participants) | 0 | 1
  SF in Toddler: Change up to 20 months |  | 0.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  SF in Young child: Change up to 20 months: number analyzed (Participants) | 0 | 1
  SF in Young child: Change up to 20 months |  | -35.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  SF in Child: Change up to 20 months: number analyzed (Participants) | 2 | 1
  SF in Child: Change up to 20 months | -20.00 (0.000) | -40.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  SF in Teens: Change up to 20 months: number analyzed (Participants) | 3 | 5
  SF in Teens: Change up to 20 months | 1.67 (7.638) | 8.00 (11.511)
  ScF in Toddler: Change up to 20 months: number analyzed (Participants) | 0 | 1
  ScF in Toddler: Change up to 20 months |  | 25.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  ScF in Young child: Change up to 20 months: number analyzed (Participants) | 0 | 1
  ScF in Young child: Change up to 20 months |  | -45.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  ScF in Child: Change up to 20 months: number analyzed (Participants) | 2 | 1
  ScF in Child: Change up to 20 months | -12.50 (10.607) | -65.00 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  ScF in Teens: Change up to 20 months: number analyzed (Participants) | 3 | 5
  ScF in Teens: Change up to 20 months | 1.67 (7.638) | -17.00 (24.135)

40. Secondary Outcome: HRQoL: Change From Baseline in EuroQoL (Quality of Life)-5 Dimensions (EQ-5D)
Description: EQ-5D considered five attributes of quality of life evaluation, that is, mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension had five possible levels: 1 (no problems); 2 (slight problems); 3 (moderate problems); 4 (severe problems), and; 5 (extreme problems). The participants rating of their current HRQoL state was recorded using a standard vertical 20-cm visual analog scale (EQ-VAS), which ranged from 0 to 100, where 0 indicated worst imaginable health state and 100 was best imaginable health state. Baseline was defined as the last non-missing value before the initial dose of HYQVIA. A negative change from baseline indicates worse health state.
Time Frame: Baseline up to 20 months
Population: Safety analysis set included all participants in the full analysis set (enrolled set) who received at least one dose of HyQvia. Here, "Overall number of Participants Analyzed" signifies participants who are evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 5 | 7
Score on a scale | -8.60 (11.149) | -4.43 (15.447)

41. Secondary Outcome: HR QoL: Change From Baseline in Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9)
Description: TSQM-9 is a 9-item, validated, self-administered instrument to assess participants satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1)*3 items = 18 for the effectiveness and convenience, and (5-1)*3 items = 12 for global satisfaction . The item scores of each of the 3 domains are summed and transformed to create a score of 0 (extremely dissatisfied) to 100 (extremely satisfied). Higher score indicated greater satisfaction in that domain. A negative change from baseline indicates less satisfaction in that domain. Baseline was defined as the last non-missing value before the initial dose of HYQVIA.
Time Frame: Baseline up to 20 months
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
Number analyzed (Participants) | 3 | 6
Score on a scale
  Effectiveness: Change at 20 months | 12.96 (32.552) | -0.92 (10.783)
  Convenience: Change at 20 months | 14.81 (27.398) | 4.63 (15.873)
  Global satisfaction: Change 20 months | 11.90 (10.911) | -2.38 (19.518)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of the study (up to 43 months)
Arm/Group | HyQvia New Starters | HyQvia Pre-treated
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/23 | 5/19
Other Adverse Events (participants affected / at risk) | 22/23 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HyQvia New Starters (N=23) | HyQvia Pre-treated (N=19)
Idiopathic orbital inflammation (Eye disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HyQvia New Starters (N=23) | HyQvia Pre-treated (N=19)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (5)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (2)
Application site pruritus (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (2)
Infusion site erythema (General disorders) | 2 (2) | 0 (0)
Infusion site pain (General disorders) | 6 (11) | 1 (1)
Infusion site pruritus (General disorders) | 4 (6) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 3 (7)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (7) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 3 (4) | 6 (12)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 3 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 6 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Solar urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT03116347/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03116347/SAP_001.pdf